CLINICAL TRIAL: NCT06024616
Title: The Impact of Group-based Life Skills and Health Empowerment for Young, Married, Women to Avoid Unintended Pregnancies in India
Brief Title: Group-based Life Skills and Health Empowerment for Married Women to Avoid Unintended Pregnancies in India
Acronym: TARANG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Network for Engineering and Economics Research and Management (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Vikalp Sansthan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD108252 (NIH); R01HD108252 (NIH)
Record Dates: First submitted 2023-08-28; First posted 2023-09-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy, Unplanned; Contraceptive Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TARANG arm (Experimental): Participants will participate in TARANG and receive the following a total of 14 sessions:
  1. Navigating newly formed relationships (e.g. spousal communication, healthy relationships with in-laws, establishing peer network, and negotiation skills)
  2. Improving women's awareness of sexual reproductive health
  3. Challenging inequitable gender norms to reduce unintended pregnancies.
  4. Life skills education to enable them to have improved social mobility, decision-making, and agency.
  The TARANG intervention will be delivered by Vikalp (a registered non-governmental organization implementing the intervention).
  Interventions: Behavioral: TARANG
- Control arm (No Intervention): Participants in the control arm receive standard of care--contraceptive access through community health workers and routine counseling by community health workers

INTERVENTIONS:
Behavioral: TARANG — TARANG is aimed to empower young women to navigate newly formed relationships, improve women's awareness of sexual reproductive health, and challenge inequitable gender norms, with an aim to reduce unintended pregnancies and increase use of family planning. The TARANG intervention for newly married women will include 14 group sessions delivered by trained moderators from Vikalp. It will cover three overarching themes, including norms, empowerment, and sexual and reproductive health and wellbeing.
  Four light-touch sessions for mothers-in-law and one in-person session for husbands of newly married women will be conducted. For husbands, TARANG will include one 2-hour group session within the first month of the intervention, followed by regular and moderated content delivery via videos and take-home exercises over WhatsApp groups. Vikalp will conduct door-to-door listing, and a research team from NEERMAN will recruit households into the study depending on the eligibility criteria.
  Arms: TARANG arm

SUMMARY:
The goal of the cluster randomized trial is to evaluate the impact of a reproductive health and empowerment intervention (TARANG) compared to the standard of care health information (control group) on the prevalence of contraceptive use and time-to-pregnancy (primary outcomes) in Rajasthan, India.

Participants will participate in TARANG intervention and receive the following sessions:

1. Navigating newly formed relationships (e.g. spousal communication, healthy relationships with in-laws, establishing peer network, and negotiation skills)
2. Improving women's awareness of sexual reproductive health
3. Challenging inequitable gender norms with an aim to reduce unintended pregnancies.
4. Life skills education to enable them to have improved social mobility, decision-making, and agency.

Investigators will compare the TARANG intervention with the standard of care to see if it delays unintended pregnancies among women.

ELIGIBILITY:
Inclusion Criteria for newly married women:

* Age 18-25 years at the time of the wedding
* Married women have permanently moved in their husbands home in the most recent wedding season (recruitment month going backwards up to October of the previous year)
* Not wanting to get pregnant within 1 year at recruitment/enrollment
* Have not had a live birth previously and not currently pregnant
* Women not planning to migrate out of the area for the period of the intervention

  • Has a living husband who is willing to consent and participate in the study in person or remotely (over phone)
* Has a living, co-residing mother-in-law type person* (see definition below) who is willing to consent and participate in the study in person (A mother-in-law type of person should be staying in the same household for the period of the intervention and has consented to participate in the study. Mother-in-law is defined as any senior woman (from a previous generation of the DIL) who are responsible for their daughter-in-law and cohabiting in the same household as their daughter-in-law (Note - household would mean a family unit which shares the same kitchen). This will usually be the biological mother of the husband, but it can be stepmother, grandmother, aunt, etc.)

Inclusion criteria for husband:

* 18 years or more at the time of the wedding
* Mother and wife are eligible for the study participation

Inclusion criteria for mother-in-law:

* Consent to participate in the study
* Assents for daughter-in-law to participate in the study
* Son and the daughter-in-law are eligible for study participation

Exclusion criteria for newly married women:

* Wanting to have a child in the next 12 months at the time of baseline
* Cognitive ability to participate in surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of unintended pregnancy | 6 months and 18-months follow-up
  Data for analysis consist of time 'at risk' - active in the study and not known to be pregnant already - and the binary outcome of 'unintended' pregnancy. The binary outcome of pregnancy will be as per self-reported answers during Demographic Health Survey style monthly calendar on whether pregnant at any time during the month, and whether the pregnancy was planned / wanted. Since eligibility is based on participants stating that they wanted to wait at least a year to get pregnant, that it was "up to god" or they didn't know, the primary outcome will assume that all pregnancies were unintended. Additional sensitivity analyses will be done with a second definition of "unintended pregnancy" to accommodate intention to change over time, so only pregnancies where respondents said they wanted to delay in the prior round will be counted as unintended.
Modern contraceptive use | 6 months and 18-months follow-up
  This will be calculated at the endline (18-months post survey) based on women's self-reported data through a detailed set of questions modeled on the Demographic Health Survey's contraceptive calendar question. For each month of the study/follow-up period, women will be asked whether they used any contraceptive method, and if yes, which type(s). A binary indicator of modern contraceptive use by month will be constructed. Modern contraceptive methods will include copper-T (intrauterine device), (Antara) injectable, emergency contraception, oral contraceptive pill, male and female condoms, male and female sterilization, lactational amenorrhea method, foam/jelly, diaphragm and standard-days method), as defined by the Demographic Health Survey in India. Person months during pregnancy and immediate postpartum will be censored for this analysis.

SECONDARY OUTCOMES:
Desired pregnancy | 6 months and 18-months follow-up
  Continuous outcome. Stated pregnancy intention using an adapted Desire to Avoid Pregnancy (DAP) Scale. Self-assessed preferences for having a baby will be measured using the DAP Scale. The DAP scale is a 14-item measure of a person's preferences about a future pregnancy and childbearing. Each item is scored from 0-4, with higher scores indicating a greater preference to avoid pregnancy but investigators will use the 9-items on childbirth given the needs of the target population.
Individual attitudes towards intimate partner violence (IPV) | 6 months and 18-months follow-up
  7-item scale that measures attitudes towards intimate partner violence against women. To construct the index, items are summed to create a score ranging from 0-7. This has been validated in India (in the Demographic Health Surveys). To be used as a continuous outcome.
Measures of reproductive autonomy/empowerment | 6 months and 18-months follow-up
  The Women's and Girls' Sexual and Reproductive Health (SRH) Empowerment Index was adapted to have 26 relevant items for existence of choice (autonomy) sub-scales and exercise of choice (self-efficacy (SE), decision-making (DM), negotiation (NG)) subscales. To construct the index, summary scores for each domain and outcome by averaging scores for relevant items are computed. Three outcome-specific empowerment scores (sexual empowerment, contraceptive empowerment and pregnancy empowerment) can be computed by adding the relevant summary scores for the existence of choice and exercise of choice domains. Finally, to examine the contribution of empowerment across the three SRH dimensions, a multidimensional SRH additive index comprising all items included in the three empowerment subscales can be computed. To be used as continuous outcome.
Time to pregnancy | 6 months and 18-months follow-up
  Continuous outcome. This will be calculated as time elapsed in months between the date of study enrollment and date of last missed period constructed on basis of documentary records or recall. This will be constructed for intended/unintended, terminated/aborted, and full term pregnancies as reported by the woman.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Vikalp Sansthan, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project and completion of the planned statistical analyses, UCSF and NEERMAN will create a de-identified dataset to be hosted on a public data-sharing platform per the guidance of the latest NIH data sharing. Until then, in accordance with this data-sharing agreement, co-investigators on the research team will not share the dataset with outsiders unless these individuals have signed a data-sharing agreement and this agreement is approved by the Principal and site co-investigators on the research team.
Supporting Information: Study Protocol
Time Frame: At the end of 2027 when the main study ends, investigators will share a de-identified dataset to be hosted on OpenICPSR, a portal approved by NIH for sharing data. It will be available indefinitely.

REFERENCES:
- [Derived] Diamond-Smith N, Gopalakrishnan L, Leslie H, Katz E, Harper C, Weiser S, Patil SR. Life skills and reproductive health empowerment intervention for newly married women and their families to reduce unintended pregnancy in India: protocol for the TARANG cluster randomised controlled trial. BMJ Open. 2024 Apr 30;14(4):e086778. doi: 10.1136/bmjopen-2024-086778. PMID 38688674